CLINICAL TRIAL: NCT03618069
Title: Diagnosis by Comprehensive Cardiovascular Imaging for Stroke and Transient Ischaemic Attacks
Brief Title: Diagnosis by Comprehensive Cardiovascular Imaging for Stroke and TIA
Acronym: DCCIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GN17ST585
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Stroke; Transient Ischaemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine investigation (No Intervention)
- study protocol CCI (CTA, cardiac CT) and MRI scans (Active Comparator)
  Interventions: Diagnostic Test: CCI scanning (CTA, cardiac CT), and MRI scanning

INTERVENTIONS:
Diagnostic Test: CCI scanning (CTA, cardiac CT), and MRI scanning — Scanning
  Arms: study protocol CCI (CTA, cardiac CT) and MRI scans

SUMMARY:
Stroke affects over 125,000 people each year in the UK and leaves at least 50% disabled. After a first stroke, there is a significant risk of recurrence (around 5-10% over the first year). While there are benefits from addressing general risk factors such as exercise, weight and smoking, selecting the best treatments for preventing a further stroke depends on understanding the underlying mechanism. Most strokes results from a blood clot causing a blockage in a blood vessel in the brain ("ischaemic" strokes, about 85% of cases). The clot may originate in the heart, the major blood vessels supplying the head, or result from disease of the small blood vessels in the brain itself (around 25% of cases each), and in around 25% of people a cause cannot be determined (sometimes because more than one exists). Different treatments are given depending on cause (for example, anticoagulant medication for clots from the heart, surgery for some arising from large arteries in the neck).

Current investigations involve multiple tests spread across different hospital departments, and commonly take several weeks to be completed. This may contribute to a high rate of strokes of uncertain cause, and may delay the start of the best treatment.

This trial will investigate the value of a single comprehensive scan to look at the heart and major blood vessels (using CT scanning) in a pilot study, comparing the classification of causes of stroke and the time to starting treatments with routine care, in a randomised study of patients with recent stroke or transient ischaemic attack (TIA, a short-lived stroke episode).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischaemic stroke or TIA
* Male or non-pregnant female≥18 years of age.
* Informed consent.

Exclusion Criteria:

* Known impaired renal function precluding contrast Computed Tomography (CT).
* Contraindications to MRI scans
* Known severe hypersensitivity to iodine based contrast media for CT or gadolinium based contrast agents for MRI.
* Severe concurrent medical condition that would prevent participation in study procedures (e.g. severe pulmonary oedema or severe septicemia) or with life expectancy ≤ 1 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with stroke of uncertain aetiology by ASCO system classification by day 30. Uncertain aetiology may include cases where insufficient investigation prevents aetiological classification. | 30 days

SECONDARY OUTCOMES:
Time to reach final aetiological classification | 30 days
Medication usage | 30 days
Diagnostic investigation usage | 30 days
Incidence of new stroke or TIA | 30 days

IPD SHARING:
Plan to Share IPD: Undecided